CLINICAL TRIAL: NCT02092194
Title: Effectiveness of High-volume Online Hemodiafiltration Compared to Standard Volume Online Hemodiafiltration. A Prospective, Multicenter, Randomized, Open-labelled Interventional Study.
Brief Title: High Versus Standard Volume Hemodiafiltration in Asia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Hemodialysis Study Group (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Sung Gyun Kim, Professor, Korean Hemodialysis Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHSG-201301
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: End-stage Renal Disease
Keywords: beta 2-Microglobulin; Hemodiafiltration; convective volume
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Dose online HDF (Active Comparator): Proposed target convection volume; 16.8-21.5 L/treatment (70-90 mL/min)
  Interventions: Procedure: Standard Dose Online HDF
- High Dose online HDF (Experimental): Proposed target convection volume; 33-43 L/treatment (140-180 mL/min).
  Interventions: Procedure: High Dose Online HDF

INTERVENTIONS:
Procedure: High Dose Online HDF — Convection volume; 33-43 L/treatment (140-180 mL/min)
  Other Names: High Volume online hemodiafiltration
  Arms: High Dose online HDF
Procedure: Standard Dose Online HDF — convection volume; 16.8-21.5 L/treatment (70-90 mL/min)
  Other Names: Standard Volume online hemodiafiltration
  Arms: Standard Dose online HDF

SUMMARY:
Online hemodiafiltration (HDF) may improve clinical outcome in end-stage renal disease. The supported mechanism is the improved clearance of uremic toxins by convective transporter. However, It has not been elucidated which convection volume is optimal, especially in Asia. A total of 60 participants receiving conventional hemodialysis will be randomly assigned to receive either high dose convective volume (33-43 L/treatment) post-dilution online HDF or standard dose (16.8-21.5 L/treatment) for 24 weeks. The primary outcome is the change of serum β2 microglobulin levels between baseline and after 24 weeks. The secondary outcomes will include changes in the nutritional markers, inflammatory markers, and blood pressure from baseline to after treatment.

This would be the first multicenter prospective, randomized controlled trial to determine whether large convective volume improves the treatment efficacy in Korean patients undergoing post-dilution online HDF.

ELIGIBILITY:
Inclusion Criteria:

* Patients on thrice-weekly standard hemodialysis for > 3 months
* Patients with a vascular access capable of delivering consistently a high blood flow rates ( ≥ 300 mL/min)
* Patients willing to provide written informed consent.

Exclusion Criteria:

* Patients with active infectious or uncontrolled inflammatory disorders
* Patients with any uncontrolled malignant disease
* Patients with recent major cardiovascular disease during the last 6 months
* Patients who are likely to receive kidney transplant within the following 1 year
* Patients whose life expectancy < 12 months
* Patients considered by investigator to have difficulty in participation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
changes in the serum concentration of β2 microglobulin | between baseline and 24 weeks after treatment

SECONDARY OUTCOMES:
Dialysis Adequacy | 24 weeks
  Kt/V by the single pool variable volume formula.
Inflammatory markers | 24 weeks
  C-reactive protein (CRP), interleukin-6, tumor necrosis factor-α.
Nutritional status | 24 weeks
  normalized protein nitrogen appearance rate, serum albumin, serum protein, subjective global assessment (SGA)
Intradialytic hypotension | 24 weeks
  Number of episode of symptomatic hypotension
Quality of Life | baseline and 24 weeks after treatment
  SF-36-K (Korean version)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Yong Cho, MD, Study Director — Korea University
Locations (6):
- South Korea (6):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Shamyook Medical Center, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul